CLINICAL TRIAL: NCT04261153
Title: Use of Cognitive Stimulation Software for Patients Over the Age of 70 Followed for Breast Cancer: COG-TAB-AGE Feasibility Study
Acronym: COG-TAB-AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A03112-55
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Cognition
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitive stimulation (Other): 3 cognitive stimulation sessions in total from the HAPPYNeuron® software, approximately 20 minutes each and spread over several days
  Interventions: Other: Cognitive stimulation

INTERVENTIONS:
Other: Cognitive stimulation — 3 cognitive stimulation sessions in total from the HAPPYNeuron® software, approximately 20 minutes each and spread over several days

SUMMARY:
Numerous studies have shown the impact of anti-cancer treatments on cognition and more particularly that of chemotherapy. Elderly patients also seem to be at higher risk of developing cognitive impairment. These disorders can have a particularly negative impact in this population, in particular by having repercussions on the observance of oral treatments or even on autonomy. However, investigators still have little data concerning the management of cognitive disorders induced by oncology treatments, particularly in the elderly patient. It is therefore necessary to offer care adapted to this population which will allow the reduction of the sequelae induced by cancer treatments and the improvement of the quality of life of elderly patients.Although there are no preventive measures yet, recent studies of young women being treated for breast cancer with a cognitive complaint have shown a beneficial effect of cognitive stimulation on these cognitive disorders. Stimulation programs of this type have been developed in electronic format. However, to date, they have not been the subject of specific studies with elderly patients in whom the use of computer interface can be an obstacle.Sponsor propose to set up a study aimed at evaluating the feasibility of using cognitive stimulation software on tablets with elderly patients.The HAPPYNeuron® software, developed by a French team of neurologists, speech-language pathologists and psychiatrists, offers exercises to be performed online to stimulate the cognitive functions most impaired by oncological treatments (memory, attention, executive functions and speed of treatment).For this feasibility study, the sponsor plan to include 50 patients aged 70 and over to have them test the acceptance of cognitive stimulation by this software with a tablet interface.

ELIGIBILITY:
Inclusion Criteria:

* Patient with breast cancer, aged 70 and over,
* During treatment with chemotherapy, targeted therapy or radiotherapy.
* Whatever the stage of the disease,
* Hospitalised in a week hospital, in traditional hospitalisation for an intercurrent episode or day hospitalisation, or undergoing radiotherapy
* Absence of major cognitive impairment preventing cognitive tests (compliance with the MoCA score threshold based on the patient's age and educational level according to GRECOGVASC standards),
* Patient with education level 3 "end of primary education" minimum (Barbizet scale),
* Mastery of the French language,
* Patient who signed the consent to participate in the study.

Exclusion Criteria:

* Hospitalization for neurological reasons (e.g. confusion), or psychiatric,
* Documented brain metastases,
* History of brain radiation therapy,
* Progressive psychiatric pathology or known dementia,
* Abuse of alcohol or drug use,
* Severe visual and / or hearing loss,
* Patient's refusal to participate,
* Patient deprived of liberty or under guardianship.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Acceptance rate | between inclusion to 1 week
  Satisfaction questionnary (Patient satisfaction questionnary; minimum 1 to maximum 5; 8 questions)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Binarelli G, Lange M, Santos MD, Duivon M, Capel A, Fernette M, Boue A, Grellard JM, Tron L, Ahmed-Lecheheb D, Clarisse B, Rigal O, Le Fel J, Joly F. Digital cognitive stimulation in elderly breast cancer patients: the Cog-Tab-Age feasibility study. BMC Complement Med Ther. 2024 May 31;24(1):209. doi: 10.1186/s12906-024-04507-0. PMID 38822324